CLINICAL TRIAL: NCT06226896
Title: Effects of Dapagliflozin on Progression of Alport Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Prof., Nanjing University School of Medicine
Other Study IDs: 2023DZKY-094
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dapagliflozin + RAS inhibitor: In addition to ACEI/ARB treatment, patients will receive dapagliflozin 10mg once daily for 24 months.
  Interventions: Drug: Dapagliflozin 10mg Tab
- RAS inhibitor only: Patients will continue ACEI/ARB treatment for 24 months.

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10mg daily plus RAS inhibitor
  Other Names: Dapagliflozin
  Groups: Dapagliflozin + RAS inhibitor

SUMMARY:
Recently, a series of large clinical trials have confirmed the cardio-renal protective effects of sodium-glucose cotransporter 2 (SGLT2) inhibitors. but few patients with hereditary nephritis were included in these studies. This study is to evaluate the effects of dapagliflozin on slowing kidney disease progression in patients with Alport syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or genetic confirmation of Alport syndrome;
* eGFR ≥ 30 ml/min/1.72m2;
* Proteinuria > 0.5 g/24 h;
* Use of an ACE inhibitor or ARB, dose stable for more than 4 weeks;

Exclusion Criteria:

* Concurrence of other types of kidney disease;
* type 1 or type 2 diabetes;
* use of other types of sodium-glucose cotransporter 2 inhibitors within the month prior to enrollment, or prior allergy to such drugs;
* ACEI combined with ARB, or direct renin inhibitors, aldosterone receptor antagonists;
* Uncontrolled hypertension (blood pressure greater than 160/90 mmHg during screening);
* Patients undergoing renal transplantation or maintenance dialysis treatment;
* Coexist with other serious and/or unstable diseases, such as serious cardiovascular diseases, respiratory diseases, liver diseases or neuropsychiatric diseases;
* Patients who are participating in clinical trials of other drugs;
* Pregnant or lactating women, or patients who do not want to receive contraception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alport syndrome who are at risk for kidney disease progression
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of eGFR | 24 months
  The change of eGFR from baseline after 24 months of treatment

SECONDARY OUTCOMES:
Change of proteinuria | 24 months
  The change of proteinuria from baseline after 24 months of treatment
Progression of kidney disease | 24 months
  The incidence of doubling of serum creatinine, a sustained ≥40% eGFR decline from baseline, or end-stage kidney disease after treatment

OTHER OUTCOMES:
Change of eGFR in different subgroups | 24 months
  The change of eGFR from baseline in patients with different phenotype -genotype after treatment
Change of proteinuria in different subgroups | 24 months
  The change of proteinuria from baseline in patients with different phenotype -genotype after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yu An, MD, Principal Investigator — National Clinical Research Center of Kidney Diseases
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided